CLINICAL TRIAL: NCT04573725
Title: Early Phase 2 Clinical Study of TS-142 in Patients with Insomnia Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TS142-201
Record Dates: First submitted 2020-09-25; First posted 2020-10-05 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2020-10

CONDITIONS: Insomnia Disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — TS-142

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 5 mg (Experimental): Period in which participants received single-dose of 5 mg TS-142 prior to bedtime
  Interventions: Drug: TS-142
- 10 mg (Experimental): Period in which participants received single-dose of 10 mg TS-142 prior to bedtime
  Interventions: Drug: TS-142
- 30 mg (Experimental): Period in which participants received single-dose of 30 mg TS-142 prior to bedtime
  Interventions: Drug: TS-142
- Placebo (Placebo Comparator): Period in which participants received single placebo prior to bedtime
  Interventions: Drug: Dose-matched Placebo to TS-142

INTERVENTIONS:
Drug: TS-142 — Participants received single-dose of 5, 10, 30 mg of TS-142 (oral capsule)
  Arms: 10 mg; 30 mg; 5 mg
Drug: Dose-matched Placebo to TS-142 — Participants received single dose-matched placebo to TS-142 (oral capsule)
  Arms: Placebo

SUMMARY:
Multicenter, randomized, placebo-controlled, 4-arm, 4-period crossover double-blind comparative study.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* Patients diagnosed with insomnia disorder according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
* Patients who scored 15 or higher on the Insomnia Severity Index (ISI) at Visit 1
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Patients with a history of any of the following diseases according to the DSM-5 criteria:

  1. Hypersomnolence disorder
  2. Narcolepsy
  3. Breathing-related sleep disorders
  4. Circadian rhythm sleep-wake disorder
  5. Parasomnias
  6. Restless legs syndrome
  7. Substance/medication-induced sleep disorder
* Patients complicated with organic brain disease (including neurodegenerative disease, cerebrovascular disorder), and/or epilepsy
* Patients with a history of poorly controlled diabetes mellitus (HbA1c >8%)
* Patients with difficulty in sleeping due to medical problems such as pain, pruritus, heart disease, nocturia (>3 times per night), bronchial asthma, reflux oesophagitis, endocrine disease, hot flush, and periodic limb movement disorder
* Other protocol defined exclusion criteria could apply

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-02-13 (Actual)

PRIMARY OUTCOMES:
LS mean difference of LPS from placebo | Day 1
  LPS is defined as the duration of time from the light off to the first persistent (10 consecutive minutes) sleep episode as measured by overnight PSG.
LS mean difference of WASO from placebo | Day 1
  WASO is defined as the time spent in wakefulness from the first persistent (10 consecutive minutes) sleep episode to the light on as measured by overnight PSG.

SECONDARY OUTCOMES:
LS mean difference of TST from placebo | Day 1
  TST is defined as the time spent in sleep from the light off to the light on as measured by overnight PSG.

CONTACTS AND LOCATIONS:
Overall Officials: Toshiro Heya, Study Director — Taisho Pharmaceutical Co., Ltd.
Locations (1):
- Taisho Pharmaceutical Co., Ltd selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Uchiyama M, Kambe D, Imadera Y, Kajiyama Y, Ogo H, Uchimura N. Effects of TS-142, a novel dual orexin receptor antagonist, on sleep in patients with insomnia: a randomized, double-blind, placebo-controlled phase 2 study. Psychopharmacology (Berl). 2022 Jul;239(7):2143-2154. doi: 10.1007/s00213-022-06089-6. Epub 2022 Mar 17. PMID 35296912